CLINICAL TRIAL: NCT04356651
Title: Efficacy of Fu's Subcutaneous Needling for Knee Osteoarthritis: a Single-blind and Randomized-controlled Trial
Brief Title: Fu's Subcutaneous Needling Treatment for Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Li-Wei Chou, Minister of Rehabilitation, China Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMUH107-REC3-027
Record Dates: First submitted 2020-04-20; First posted 2020-04-22 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Knee Osteoarthritis
Keywords: Fu's subcutaneous needling; myofascial trigger point; muscle tone
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fu's subcutaneous needling(FSN) (Experimental): In this arm, the subjects will receive the intervention of FSN on Day1, Day2 and Day4, in total 3 treatments. The subjects will receive assessments before and after each interventions. After total treatments finished, the subjects will receive assessments on Day8 and Day15, separately.
  Interventions: Procedure: Fu's subcutaneous needling(FSN)
- Transcutaneous Electric Nerve Stimulation (Active Comparator): In this arm, the subjects will receive the intervention of Transcutaneous Electric Nerve Stimulation on Day1, Day2 and Day4, in the total 3 treatments. The subjects will receive assessments before and after each interventions. After total treatments finished, the subjects will receive assessments on Day8 and Day15, separately.
  Interventions: Procedure: Transcutaneous Electric Nerve Stimulation

INTERVENTIONS:
Procedure: Fu's subcutaneous needling(FSN) — In this study, physician will use a disposable Fu's subcutaneous needling(FSN) to penetrate the subject's skin from anterior superior iliac spine(ASIS) to 1/3 superior border of patella. Then the physician will push forward the needle parallel to the skin surface. The physician will sway the needle 45 times in 30 seconds. After swaying the needle, the physician will instruct the subject to do sole dorsiflexion for 10 seconds resisting the physician's opposite force, then the subject take a rest for 10 seconds. The above actions are 3 repetitions. Then the subject do knee flexion and extension for 10 seconds, and take a rest for 10 seconds. These actions are also 3 repetitions. After the above reperfusion approach of muscles, the physician will take out the needle to finish the treatment.
  Arms: Fu's subcutaneous needling(FSN)
Procedure: Transcutaneous Electric Nerve Stimulation — Transcutaneous electrical nerve stimulation (TENSor TNS) is the use of electric current produced by a device to stimulate the nerves for therapeutic purposes. TENS, by definition, covers the complete range of transcutaneously applied currents used for nerve excitation although the term is often used with a more restrictive intent, namely to describe the kind of pulses produced by portable stimulators used to treat pain. The unit is usually connected to the skin using two or more electrodes. A typical battery operated TENS unit is able to modulate pulse width,frequency and intensity. Generally TENS is applied at high frequency (>50 Hz) with an intensity below motor contraction (sensory intensity) or low frequency (<10Hz) with an intensity that produces motor contraction.
  Arms: Transcutaneous Electric Nerve Stimulation

SUMMARY:
The population affected by degenerative knee arthritis is very large. The investigator performed Fu's subcutaneous needling (FSN). This experiment used a randomized single-blind experiment to assess the immediate, short-term and long-term effects of Fu's subcutaneous needling (FSN) therapy on patellar pain in patients with degenerative arthritis.

DETAILED DESCRIPTION:
The population affected by degenerative knee arthritis is very large. According to a survey conducted by the Ministry of Health and Welfare, the prevalence of osteoarthritis of the knee in Taiwan is about 3.5 million people, accounting for about 15% of the total population. Its effects are a heavy burden on socio-economic costs, and in addition to being included in medical expenses, serious cases can lead to incapacity to work; therefore, the disease is an important factor in causing disability and disability First, it is worth our attention.

Floating needle is a kind of dry needle therapy, which has been used in the treatment of degenerative arthritis for more than 20 years. It has been clearly annotated in the treatment strategy that it uses disposable floating needle needles at the superficial subcutaneous fascia, Parallel to the muscle to sweep away, and with reperfusion activities, muscle pain caused by muscle fascia and soft tissue pain with immediate and good pain relief effect, but still lack of treatment and rigorous evaluation of the establishment.

For the reasons of the degenerative arthritis pain, the clinical observation is not entirely due to the cause of joint deformity or cartilage damage, soft tissue lesions around the knee is also a common source of pain, the use of floating needle for the diagnosis of soft tissue injury , And observed its efficacy, which is also the core of this study.

This experiment used a randomized single-blind experiment to assess the immediate, short-term and long-term effects of floating needle therapy on patellar pain in patients with degenerative arthritis. The assessment tools included the VAS, WOMAC , Lesquesne index, the Muscle Tension Changes in the Lower Extremities, and Gyko .

ELIGIBILITY:
Inclusion Criteria:

- 1.Volunteers who are older than 50 years old and can cooperate with the experiment.

2.Established diagnosis of unilateral or bilateral degenerative knee arthritis. 3.There is a local trigger point around the unilateral or bilateral knee joint which on the muscle of Vastus lateralis, Vastus medialis, Gastrocnemius, or Tibialis anterior.

Exclusion Criteria:

* 1.There are contraindications to general treatment, such as serious medical problems, recent serious trauma, or pregnant women.

  2.There has been a history of drug abuse (including excess alcohol) that affects pain assessors.

  3.Have received knee surgery. 4.People with central or peripheral nerve disease. 5.Cognitive impairment, unable to cooperate with the experimenter. 6.Patients currently receiving other treatments for knee osteoarthritis

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-07-07 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-01-10 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scales | 1 day
  The visual analogue scale or visual analog scale (VAS) is a psychometric response scale which can be used in questionnaires. This tool used to help a person rate the intensity of certain sensations and feelings, such as pain. A straight line of 100mm is actually marked with 0 mm on the far left and 100mm on the far right. Two faces are drawn on both ends. Explain to the patient that 0 mm means no pain and 100 mm means very painful. From the left end The right shift indicates more and more pain. Take a pen and let the patient draw a short line vertically on the line, representing his painful position, and record the measured cm value. In this test, if the score of the subject decreases, it can represent the treatment is helpful for the improvement of the patient's pain.
Pressure Pain Threshold | 1 day
  Pressure pain threshold (PPT) is defined as the minimum force applied which induces pain. This measure has proven to be commonly useful in evaluating tenderness symptom
Muscle tension | 1 day
  Muscle tension is the muscle's resistance to passive stretch during resting state. The measuring tool called Myotone will calculate three parameters such as tone, elasticity and stiffness automatically and get a value to represent the muscle tension. If the value decrease, it can represent the treatment is helpful for the subjective muscle relax.
GyKo | 1 day
  GyKo is an inertial measurement tool for the analysis of the movement of any body segment
WOMAC | 1 day
  The WOMAC measures five items for pain (score range 0-20), two for stiffness (score range 0-8), and 17 for functional limitation (score range 0-68).
Lequesne'Index | 1 day
  A pain scale measures a patient's pain intensity or other features.

CONTACTS AND LOCATIONS:
Overall Officials: Li-Wei Chou,, PhD, Principal Investigator — China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chiu PE, Fu Z, Sun J, Jian GW, Li TM, Chou LW. Efficacy of Fu's Subcutaneous Needling in Treating Soft Tissue Pain of Knee Osteoarthritis: A Randomized Clinical Trial. J Clin Med. 2022 Dec 2;11(23):7184. doi: 10.3390/jcm11237184. PMID 36498758
- [Derived] Chiu PE, Fu Z, Jian GW, Huang CH, Li TM, Chou LW. Evaluating Effectiveness of Fu's Subcutaneous Needling for the Pain Nature and Quality of Life in Patients with Knee Osteoarthritis: A Study Protocol of Randomized Clinical Trial. J Pain Res. 2021 Oct 9;14:3163-3172. doi: 10.2147/JPR.S333299. eCollection 2021. PMID 34675644